CLINICAL TRIAL: NCT06585267
Title: Development of a New Patient Reported Outcome Measure (PROM) to Assess Patient's Emotional Wellbeing, and Perceptions of Total Knee Replacement Surgery for the Treatment of Knee Arthritis Phase Four - Validation of Final Questionnaire This Phase is to Validate the Final Questionnaire in Terms of Reliability, Validity and Ability to Detect Change
Brief Title: Development of a New Patient Reported Outcome Measure (PROM) to Assess Patient's Emotional Wellbeing, and Perceptions of Total Knee Replacement Surgery for the Treatment of Knee Arthritis
Acronym: SYNC01- P4
Status: Active, not recruiting | Type: Observational
Sponsor: Invibio Ltd (Industry)
Collaborators: Oxford University Innovation (Unknown)
Responsible Party: Sponsor
Other Study IDs: SYNC01- P4
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Complete Questionnaires Following TKR Surgery
Keywords: TKR; Questionnaire

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main patient Group: Patients who have undergone Total Knee Replacement (TKR) Surgery

SUMMARY:
Development of a new Patient Reported Outcome Measure (PROM) to assess patient's emotional wellbeing, and perceptions of Total Knee Replacement surgery for the treatment of knee arthritis.

DETAILED DESCRIPTION:
Patients will complete the final developed questionnaire for quantitative analysis only (involves no administration of any medicinal products or medical devices) and is considered a low-risk project.

Patients will also be asked to complete the already validated EQ-5D-5L and Oxford Knee Score questionnaires at the same time as the final developed questionnaire following their Total Knee Replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years of age or older.
* Patients who have undergone Total Knee Replacement surgery with a metal implant for the treatment of end-stage knee arthritis in the last 3 months.
* Patients who have only undergone one Total Knee Replacement surgery on the index knee.
* Patients who, in the opinion of the Investigator, are able to understand this project and co-operate with the requirements of participation.
* Patients who are able to give voluntary, written informed consent to participate in this project and from whom consent has been obtained.

Exclusion Criteria:

* Patients, who in the opinion of the Investigator, exhibit evidence of any condition or co-morbidity that would compromise their participation in the project.
* Patients who are unable to understand and communicate fluently in English.
* Patients who have experienced a complication following Total Knee Replacement surgery requiring a further hospital admission or revision surgery to the index knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are due to undergo TKR surgery or have undergone TKR surgery in the last 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Validate final questionnaire | From first post-op visit to 12month follow-up
  Validation of final questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Professor Hemant Pandit, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- Chapel Allerton Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only collated validated findings will be shared no individual data will be